CLINICAL TRIAL: NCT01454648
Title: Severe Traumatic Brain Injury - Comparison of Outcome in Paramedic Versus Physician Staffed Emergency Medical Services
Brief Title: Prehospital Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R09161
Record Dates: First submitted 2011-10-05; First posted 2011-10-19 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2014-11

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; EMS; Out-of-Hospital
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Physician-staffed: Patients treated by physician-staffed emergency medical service (EMS) unit
- Paramedic-staffed: Patients treated by paramedic-staffed emergency medical service (EMS) unit

SUMMARY:
The aim of the study is to measure the effect of Finnish physician-staffed EMS unit treatment methods on traumatic brain injury (TBI) patient prognosis.

DETAILED DESCRIPTION:
A secondary aim is to identify out-of-hospital treatment factors that can be influenced by education and protocols.

ELIGIBILITY:
Inclusion Criteria:

* TBI with GCS ≤ 8 or unconsciousness verified by an on-call neurosurgeon during admission to the hospital.

Exclusion Criteria:

* Multiple trauma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2005-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 year

SECONDARY OUTCOMES:
Glasgow outcome score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arvi Yli-Hankala, professor, Study Director — Tampere University Hospital; Toni Pakkanen, M.D., Principal Investigator — Tampere University; Ilkka Virkkunen, M.D., PhD, Study Director — Tampere University Hospital; Tom Silfvast, M.D., PhD, Study Director — Helsinki University Central Hospital; Tarja Randell, M.D., PhD, Study Chair — Helsinki University Central Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Pakkanen T, Virkkunen I, Kamarainen A, Huhtala H, Silfvast T, Virta J, Randell T, Yli-Hankala A. Pre-hospital severe traumatic brain injury - comparison of outcome in paramedic versus physician staffed emergency medical services. Scand J Trauma Resusc Emerg Med. 2016 Apr 29;24:62. doi: 10.1186/s13049-016-0256-x. PMID 27130216